CLINICAL TRIAL: NCT02279693
Title: Evaluation of the Dose Received by the Prostate With in Vivo Dosimetry in Patients Treated With Daily IGRT Associated With IMRT Using Two Repositioning Techniques for Localized Prostate Cancer
Acronym: PROSTRACK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: feasibility problem
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-A00122-45
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: Raypilot dosimetry; CBCT (cone beam computed tomography)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Fiducial Markers; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBCT (Other): cone beam computed tomography (CBCT) repositioning
  Interventions: Other: CBCT; Radiation: IGRT Associated With IMRT
- fiducial markers (Other): kV imaging of fiducial marker repositioning
  Interventions: Other: fiducial marker (kV imaging); Radiation: IGRT Associated With IMRT

INTERVENTIONS:
Other: CBCT — 10 participants will receive a cone beam computed tomography (CBCT) repositioning
  Arms: CBCT
Other: fiducial marker (kV imaging) — 10 participants will receive a kV imaging of fiducial marker repositioning.
  Arms: fiducial markers
Radiation: IGRT Associated With IMRT

SUMMARY:
This study evaluates the dose received by the prostate with in vivo dosimetry when delivering image guided radiation therapy (IGRT) associated with intensity modulated radiation therapy (IMRT) for patients with localized prostate cancer using two repositioning techniques: fiduciary markers or soft tissues.

DETAILED DESCRIPTION:
10 participants will receive a cone beam computed tomography (CBCT) repositioning, while the other 10 will receive a kV imaging of fiducial marker repositioning. The principal objective is to evaluate and compare the dose received by the prostate using two repositioning techniques.

ELIGIBILITY:
Inclusion Criteria:

* male > 18 years
* carcinoma of the prostate histologically confirmed
* OMS 0-1
* localized stage
* favorable, intermediate and unfavorable groups according to NCCN or D'Amico classification
* patients must have signed a written informed consent form
* patients must be affiliated to a Social Health Insurance.

Exclusion Criteria:

* metastasis
* indication for pelvic radiation
* anticoagulant therapy
* lateral or bilateral hip replacement
* patient receiving an adult protective services
* Patient unable to comply with the required medical follow-up for geographic, social or psychological reasons

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12-22 (Actual); Primary Completion 2014-12-22 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
dosimetry (measurement of the absorbed dose, delivered to prostate, by ionizing radiation) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gilles CREHANGE, MD, PhD, Principal Investigator — Centre Georges François Leclerc
Locations (1):
- Centre Georges-François Leclerc, Dijon, France